CLINICAL TRIAL: NCT00687661
Title: The Use of Bisphosphonates to Prevent or Delay the Progression of Vascular Calcification in End-Stage Renal Disease: A Randomized Controlled Trial
Brief Title: Queen's University Investigation of Calcification in Chronic Kidney Disease
Acronym: QUICK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Karen Yeates, Dr Karen E. Yeates, Department of Medicine Queen's University., Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QUICK Study; J.P.Bickell Foundation Grant; 8 April 2005
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Failure; Vascular Calcification; Bisphosphonates
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Vascular Calcification | interventions — Diphosphonates

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Arm #1 will include patients randomized to receive bisphosphonate therapy for 24 months.
  Interventions: Drug: Bisphosphonate
- 2 (Placebo Comparator): Arm #2 will include patients randomized to receive placebo therapy for 24 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bisphosphonate — 35mg given orally once weekly for 24 months
  Other Names: Residronate
  Arms: 1
Drug: Placebo — identical placebo pill once weekly for 24 months
  Arms: 2

SUMMARY:
Kidney disease is a fundamental part of medicine because of its prominence in Western society. Common conditions such as diabetes, hypertension and kidney infections can all progress to End-Stage Renal Disease (ESRD) also known as Stage 5 chronic kidney disease (CKD 5). Once ESRD has begun, kidney function is poor at best, thus the body is unable to effectively clear harmful toxins from the blood.

A common feature of ESRD is vascular calcification, a process where blood vessels (especially arteries) attract deposits of the mineral calcium. Over time, these deposits harden and thicken in the layers of blood vessels, which limit blood flow to body tissues and can produce significant disease including hypertension, heart disease and stroke. Although the process of vascular calcification is unknown, there is mounting evidence that it is mediated by cellular events that are similar to those seen in bone formation with in the body (osteogenesis). With this point in mind, it has been suggested that agents medicine employs to limit excess bone formation will reduce the rate of vascular calcification in CKD Stage 5.

This study will employ one group of drugs called bisphosphonates which have been used to limit bone formation. It will study their effect on vascular calcification in adult dialysis patients.

DETAILED DESCRIPTION:
Presently, there exist few therapies aimed at retarding the progression of vascular calcification. One study showed that agents that limit the absorption of phosphate from food (phosphate binders) slow the progression of vascular calcification, and as a result, treatments emphasize phosphate control through diet and phosphate binders. Other studies have shown that the use of statins, to lower LDL cholesterol levels may reduce the progression of coronary calcification in non-ESRD patients, but data from ESRD are lacking. While these treatments have been helpful, the improvements in patients' outcomes have not been overwhelming positive.

This proposed study is not the first to study the use of bisphosphonates on vascular calcification. Repeated studies have shown impressive reduction in calcification rates in several animal models, which begs the question, how will bisphosphonates fare in human subjects? Preliminary research has begun, but clearly an expansive trial on humans is needed to explore the use of a promising therapy. Our study hopes to provide insight into this area of cardiovascular research.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* receiving maintenance renal replacement therapy for less than 12 months
* incident patients starting renal replacement therapy for the first time

Exclusion Criteria:

* active vasculitis
* severe hypocalcemia
* previous adverse side effect to bisphosphonate use
* current use of corticosteroids
* weight greater than 300 pounds
* pregnancy
* not expected to survive greater than one year
* expected to discontinue renal replacement therapy during the study period or recover renal function
* evidence of adynamic bone disease
* current bisphosphonate use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Absolute change in coronary artery calcification score (CaSc) from baseline to study completion. | 24 months

SECONDARY OUTCOMES:
Change in bone density score (wrist/hip) as calculated by Ct scanning method, # fractures, MI, Stroke, amputation/surgery for peripheral revascularization. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Yeates, Dr, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada